CLINICAL TRIAL: NCT03362437
Title: A Study to Evaluate the Pharmacokinetics of BMS-986177 From Form A and Form B in Healthy Participants
Brief Title: Evaluate the Pharmacokinetics of BMS-986177 From Two Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CV010-020
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Receive 200 mg BMS-986177 Form A without food
  Interventions: Drug: BMS-986177
- Treatment B (Experimental): Receive 200 mg BMS-986177 Form B without food
  Interventions: Drug: BMS-986177
- Treatment C (Experimental): Receive 200 mg BMS-986177 Form B with food
  Interventions: Drug: BMS-986177

INTERVENTIONS:
Drug: BMS-986177 — Form A
  Arms: Treatment A
Drug: BMS-986177 — Form B
  Arms: Treatment B; Treatment C

SUMMARY:
Assess the pharmacokinetics (fasting and fed), safety, and tolerability of BMS-986177 following oral dosing of Form A and Form B

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 32.0 kg/m2, inclusive
* Women must not be of childbearing potential (cannot become pregnant)

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Head injury in the last 2 years
* History of bleeding disorder including rectal bleeding (ie, hemorrhoids), spontaneous nosebleeds, etc.

Other protocol defined inclusion / exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 3 days
  Measured by plasma concentration
AUC from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to 3 days
  Measured by plasma concentration
AUC from time zero extrapolated to infinite time (AUC(INF)) | Up to 3 days
  Measured by plasma concentration

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 12 days
  Safety and tolerability as measured by incidence of AEs
Incidence of Serious Adverse Events (SAEs) | Up to 30 days
  Safety and tolerability as measured by incidence of SAEs
Number of participants with electrocardiogram abnormalities | Up to 12 days
Number of participants with physical examination abnormalities | Up to 12 days
Number of participants with clinical laboratory abnormalities | Up to 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Briston-Myers Squibb
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls